CLINICAL TRIAL: NCT00069160
Title: A Clinical Trial of the P-Glycoprotein Antagonist, Tariquidar (XR9576), in Combination With Docetaxel in Patients With Lung, Ovarian, Renal and Cervical Cancer: Analysis of the Interaction Between Tariquidar and Docetaxel
Brief Title: Tariquidar and Docetaxel to Treat Patients With Lung, Ovarian, Renal and Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Susan E. Bates, National Cancer Institute (NCI), National Institutes of Health (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030284; 03-C-0284 (Other: Clinical Center (CC), National Institutes of Health (NIH)); 030284 (Other: Clinical Center (CC), National Institutes of Health (NIH)); NCT00072202 (obsolete NCT alias)
Record Dates: First submitted 2003-09-15; First posted 2003-09-16 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-09

CONDITIONS: Lung Neoplasms; Ovarian Neoplasms; Cervix Neoplasms; Renal Neoplasms
Keywords: Pharmacokinetics; Pharmacodynamics; Multidrug Resistance Reversal; Molecular Target; P-Glycoprotein Inhibition; Lung Cancer; Ovarian Cancer; Cervical Cancer; Renal Cancer
MeSH Terms: conditions — Lung Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Kidney Neoplasms | interventions — Docetaxel; tariquidar; Technetium Tc 99m Sestamibi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pts who received docetaxel on day 1, 8, & tariquidar day 8,22 (Experimental): Patients receive 40 mg/m^2 docetaxel intravenous (IV) over 1 hour on days 1 and 8 and 150 mg tariquidar intravenous (IV) over 30 minutes on days 8 and 22. From cycle 2 and onward 75 mg/m^2 docetaxel was administered every 21 days in combination with a single 150 mg dose.
  Interventions: Drug: docetaxel; Drug: tariquidar; Other: 99mTc-sestamibi imaging
- Pts who received docetaxel on days 1, 8, & tariquidar day 1,22 (Experimental): Patients receive docetaxel intravenous (IV) over 1 hour on days 1 and 8 and tariquidar intravenous (IV) over 30 minutes on days 1 and 22.
  Interventions: Drug: docetaxel; Drug: tariquidar; Other: 99mTc-sestamibi imaging

INTERVENTIONS:
Drug: docetaxel — Patients receive docetaxel intravenous (IV) over 1 hour on days 1 and 8.
  Other Names: Taxotere
Drug: tariquidar — Patients receive tariquidar intravenous (IV) over 30 minutes on days 8 and 22.
  Other Names: XR9576
Other: 99mTc-sestamibi imaging — Bolus injection of 29 mCi of 99mTc-sestamibi intravenously for each imaging study.
  Other Names: Cardiolite

SUMMARY:
The purpose of this study is three-fold: 1) to examine the ability of the experimental drug tariquidar to improve chemotherapy results by blocking a protein (P-glycoprotein) on some cancer cells that acts to pump out cancer drugs; 2) examine how tariquidar interacts with the cancer drug docetaxel; and 3) evaluate the effectiveness of combination treatment with tariquidar and docetaxel in treating patients with lung, ovarian, or cervical cancer.

Patients 18 years of age and older with recurrent or metastatic (spreading) lung, cervical, or ovarian cancer who cannot benefit from any standard treatment may be eligible for this study. Candidates will be screened with a medical history and physical examination; review of pathology slides; blood and urine tests; imaging tests, including computed tomography (CT) or magnetic resonance imaging (MRI) scans; chest x-ray, electrocardiogram (EKG); and possibly echocardiogram.

Participants will undergo the following tests and procedures:

Blood draw. Blood is drawn before treatment begins to establish baseline levels for future blood tests. Blood counts are done twice weekly after chemotherapy begins.

Central venous catheter placement. A plastic tube is put into a major vein in the chest. It is used to give the study drugs or other medications, including antibiotics and blood transfusions, if needed, and to withdraw blood samples. The line is usually placed under local anesthesia in the radiology department or the operating room. It can stay in the body for months or be removed after each treatment is completed.

Chemotherapy. Treatment cycles are 21 days. Both drugs are given on day 1 of each cycle. First, tariquidar is given as a 30-minute infusion. One hour after the tariquidar infusion, docetaxel is infused over 1 hour. (For the first cycle only, docetaxel is given in divided doses one week apart and tariquidar is administered on either day 1 or day 8. The order of tariquidar administration is randomized to generate optimal pharmacokinetic data. Patients will be hospitalized for several days during this cycle to gather research data). The tariquidar dose remains the same throughout the study. Docetaxel may be increased or decreased from cycle to cycle, based on side effects.

DETAILED DESCRIPTION:
Intrinsic and acquired drug resistance remain major obstacles in the treatment of cancer. Accumulating evidence indicates that in some malignancies P-glycoprotein (Pgp) can confer resistance, and that its reversal can improve therapeutic outcome. Clinical trials investigating Pgp antagonists have been hampered by the occurrence of unpredictable pharmacokinetic interactions, which have required dose reductions of the chemotherapeutic agents to avert excessive toxicity. Tariquidar (XR9576) is a new Pgp antagonist that is more potent and has prolonged activity. Phase I trials with paclitaxel, vinorelbine, and docetaxel have demonstrated that tariquidar (XR9576) has minimal pharmacokinetic interactions while surrogate studies have confirmed in vivo inhibition of Pgp-mediated drug transport.This study seeks to determine the pharmacokinetic interaction, if any between docetaxel and tariquidar and to evaluate the potential for activity in lung, ovarian, primary peritoneal, fallopian tube and cervical cancers. Renal cell cancer has been added in a 3/1/06 amendment. The secondary goal is to evaluate the impact of tariquidar on uptake of (99m)Tc-sestamibi in recurrent or metastatic tumors of patients with lung, ovarian, renal or cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must fulfill all of the following criteria to be eligible for study admission:
* Age greater than or equal to 18 years.
* Histologic or cytologic confirmation of lung, cervical, or ovarian cancer, following at least one standard treatment regimen, and for which there is no known standard therapy capable of extending life expectancy. Female patients with primary papillary carcinoma of the peritoneum and fallopian tube cancers will be included in the latter group, as the disease entities are closely associated with epithelial ovarian carcinoma, can be difficult to distinguish, have a similar epithelial origin, and are treated in an identical manner.
* Histologic or cytologic confirmation of renal cell carcinoma (clear cell, type 1 and type II papillary chromophobe, collecting duct and medullary). Patients should have received either sunitinib or sorafenib, unless deemed ineligible for treatment with either agent. In addition,patient should either: (a) have received IL-2; (b) have been evaluated for therapy with Interleukin-2 (IL- 2) and deemed to be ineligible; or (c) have been evaluated for therapy with IL2 and refused treatment.
* Performance status: Eastern Cooperative Oncology Group (ECOG) 0-2
* Life expectancy of 3 months or greater.
* Suitable candidate for receiving planned therapy as evidenced by screening laboratory assessments hematologic, renal hepatic, and metabolic functions, platelet count greater than or equal to 90,000/mL, absolute granulocyte count(AGC) greater than or equal to 1,500/mL, serum creatinine greater than or equal to 1,500/mL, serum creatine less than or equal to 1.5 mg/dl )or if greater than 1.5 a measured 24 hour creatinine clearance greater than or equal to 50 mL/min) and serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 2.5 x normal limit (NL) and bilirubin less than or equal to 1.5 x NL (in patients with clinical evidence of Gilbert's disease,less than or equal to 3 x NL).
* Patients must be greater than or equal to 4 weeks prior radiation or chemotherapy, greater than 2 weeks from hormonal therapy; greater than 4 weeks from prior experimental therapy; greater than 6 weeks from mitomycin C; and greater than 8 weeks from prior UCN01 treatment.
* No serious intercurrent medical illness.
* Measurable disease by radiographic means or physical examination. For ovarian cancer, assessable disease by cancer antigen 125 (CA125) measurement is allowed.
* Willingness to sign a written consent form, and to comply with the protocol.

Exclusion Criteria:

* The following patient populations are not eligible for this study.
* Pregnant or nursing women are not eligible; women of childbearing age must agree to use an effective method of contraception. Pregnant women are not eligible because of teratogenic effects of chemotherapy.
* The presence of a second malignancy that has not received primary treatment or would complicate the primary objective of this study.
* Patients who are poor medical risk because of active, uncontrolled infection or other nonmalignant systemic disease.
* Human immunodeficiency virus (HIV) seropositive patients. Patients infected with the HIV virus will be excluded from this trial because the effect of the combination of tariquidar and docetaxel on HIV replication and/or the immune system is unknown and potentially harmful.
* Patients receiving agents which have major interactions with the cytochrome P450 3A4 (CYP3A4)drug metabolizing system and which cannot be discontinued may not be included in the trial.
* Untreated brain metastases (or local treatment of brain metastases within the last 6 months) due to the poor prognosis of these patients and difficulty ascertaining the cause of neurologic toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2003-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Bates, M.D., Principal Investigator — NCI, NIH
Locations (1):
- National Institutes of Health, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ling V, Thompson LH. Reduced permeability in CHO cells as a mechanism of resistance to colchicine. J Cell Physiol. 1974 Feb;83(1):103-16. doi: 10.1002/jcp.1040830114. No abstract available. PMID 4855907
- [Background] Akiyama S, Fojo A, Hanover JA, Pastan I, Gottesman MM. Isolation and genetic characterization of human KB cell lines resistant to multiple drugs. Somat Cell Mol Genet. 1985 Mar;11(2):117-26. doi: 10.1007/BF01534700. PMID 3856953
- [Background] Beck WT, Cirtain MC, Lefko JL. Energy-dependent reduced drug binding as a mechanism of Vinca alkaloid resistance in human leukemic lymphoblasts. Mol Pharmacol. 1983 Nov;24(3):485-92. PMID 6579344
- [Result] Kelly RJ, Draper D, Chen CC, Robey RW, Figg WD, Piekarz RL, Chen X, Gardner ER, Balis FM, Venkatesan AM, Steinberg SM, Fojo T, Bates SE. A pharmacodynamic study of docetaxel in combination with the P-glycoprotein antagonist tariquidar (XR9576) in patients with lung, ovarian, and cervical cancer. Clin Cancer Res. 2011 Feb 1;17(3):569-80. doi: 10.1158/1078-0432.CCR-10-1725. Epub 2010 Nov 16. PMID 21081657
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Groups:
- Pts Who Received Docetaxel on Day 1, 8, & Tariquidar Day 8,22: Patients receive 40 mg/m^2 docetaxel intravenous (IV) over 1 hour on days 1 and 8 and 150 mg tariquidar intravenous (IV) over 30 minutes on days 8 and 22. From cycle 2 and onward 75 mg/m^2 docetaxel was administered every 21 days in combination with a single 150 mg tariquidar dose.
- Pts Who Received Docetaxel on Days 1, 8, & Tariquidar Day 1,22: Patients receive docetaxel intravenous (IV) over 1 hour on days 1 and 8 and tariquidar intravenous (IV) over 30 minutes on days 1 and 22.From cycle 2 and onward 75 mg/m^2 docetaxel was administered every 21 days in combination with a single 150 mg tariquidar dose.
Period: Overall Study
Arm/Group | Pts Who Received Docetaxel on Day 1, 8, & Tariquidar Day 8,22 | Pts Who Received Docetaxel on Days 1, 8, & Tariquidar Day 1,22
Started | 23 | 25
Completed | 23 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pts Who Received Docetaxel on Day 1, 8, & Tariquidar Day 8,22 | Pts Who Received Docetaxel on Days 1, 8, & Tariquidar Day 1,22 | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 4 | 5 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 50.76 (9.54) | 55.77 (9.57) | 53.37 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean of Maximum Concentration of the Drug (Cmax)
Description: In the first cycle patients were to receive docetaxel on days 1 and 8 and to be randomized to receive tariquidar on either day 1 or 8. Thus pharmacokinetic data with and without tariquidar can be compared.
Time Frame: 24 hours
Population: Docetaxel alone (C1D1 = 21 patients; C1D8 = 18 patients) Docetaxel with Tariquidar (C1D1 = 21 patients; C1D8 = 16 patients) Data were evaluable in 39 patients. Paired data from 31 participants were evaluable.
Measure: Geometric Mean (95% Confidence Interval); unit: Cmax (ng/mL)
Groups:
- Docetaxel Alone: 40 mg/m^2 docetaxel over 1 hour on days 1 and 8.
- With Tariquidar: 40 mg/m^2 docetaxel intravenous (IV) over 1 hour on days 1 and 8 and 150 mg tariquidar intravenous (IV) over 30 minutes on either day 1 or 8 and then again on day 22. From cycle 2 and onward 75 mg/m^2 docetaxel was administered every 21 days in combination with a single 150 mg dose of tariquidar.
Arm/Group | Docetaxel Alone | With Tariquidar
Number analyzed (Participants) | 39 | 37
Cmax (ng/mL)
  C1D1 | 1315 [1081 to 1598] | 1093 [791.2 to 1510]
  C1D8 | 1060 [773.5 to 1452] | 1026 [807.3 to 1303]
  Both Groups (C1D1 + C1D8) | 1190 [999.9 to 1416] | 1063 [869.2 to 1301]

2. Primary Outcome: The Number of Participants With Adverse Events.
Description: Here are the total number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 4 yrs 8-11 months
Measure: Number; unit: participants
Groups:
- Patients on Docetaxel on Days 1, 8 & Tariquidar on Day 8, 22; Patients on Docetaxel on Days 1, 8 & Tariquidar on Days 1, 22: Patients receive 40 mg/m^2 docetaxel intravenous (IV) over 1 hour on days 1 and 8 and 150 mg tariquidar intravenous (IV) over 30 minutes on days 8 and 22. From cycle 2 and onward 75 mg/m^2 docetaxel was administered every 21 days in combination with a single 150 mg dose.
Arm/Group | Patients on Docetaxel on Days 1, 8 & Tariquidar on Day 8, 22 | Patients on Docetaxel on Days 1, 8 & Tariquidar on Days 1, 22
Number analyzed (Participants) | 23 | 25
participants | 23 | 25

3. Primary Outcome: Geometric Mean of Area Under Curve (AUC0)-24
Time Frame: 24 hours
Population: Docetaxel alone (C1D1 = 21 patients; C1D8 = 18 patients) Docetaxel with Tariquidar (C1D1 = 21 patients; C1D8 = 16 patients) Pharmacokinetic data were evaluable in 39 patients. Paired data from 31 participants were evaluable.
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Docetaxel Alone | With Tariquidar
Number analyzed (Participants) | 39 | 37
h*ng/mL
  C1D1 | 1367 [1126 to 1658] | 1409 [1172 to 1694]
  C1D8 | 1308 [989.8 to 1730] | 1327 [1084 to 1623]
  Both Groups (C1D1 + C1D8) | 1339 [1144 to 1568] | 1373 [1206 to 1563]
Statistical Analysis 1: Comparison: Docetaxel Alone vs With Tariquidar; Test type: Superiority or Other; p > .05, t-test, 2 sided

4. Primary Outcome: Clinical Response Rate
Description: Response is determined by RECIST criteria defined as changes in only the largest diameter (unidimensional measurement) of the tumor lesion. Lesions are either measurable or non-measurable. Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as >/- 20 mm with conventional techniques (CT, MRI, xray) or as >/- 10 mm with a spiral CT scan. Non-measurable lesions are defined as all other lesions (or sites of disease) including small lesions (longest diameter <20 mm with conventional techniques or <10 mm using spiral CT.
Time Frame: 4 years, 8-11 months
Measure: Number; unit: Percentage of participants
Groups:
- All Patients Who Received Docetaxel and Tariquidar: Patients receive 40 mg/m^2 docetaxel intravenous (IV) over 1 hour on days 1 and 8 and 150 mg tariquidar intravenous (IV) over 30 minutes on days 8 and 22. From cycle 2 and onward 75 mg/m^2 docetaxel was administered every 21 days in combination with a single 150 mg dose.
Arm/Group | All Patients Who Received Docetaxel and Tariquidar
Number analyzed (Participants) | 48
Percentage of participants | 8

5. Secondary Outcome: Percent Increase in Sestamibi Area Under Curve (AUC) in Liver After Tariquidar
Description: A significant change in the area under the curve(AUC) in liver tissue (normal tissue as a surrogate) is defined as P<0.001. A secondary objective of this study was to establish whether tariquidar (150 mg) modulates Pgp in liver. Sestamibi is a Pgp substrate that may be a surrogate for measuring drug efflux from tumors. A baseline Tc-sestamibi scan was obtained before the administration of tariquidar. A minimum of 48 hours later, on or about day 22 a single dose of tariquidar was administered, followed by a second Tc-sestamibi scan.
Time Frame: 3 - 24 hours
Population: Percent increase in sestamibi AUC in liver after tariquidar.
Measure: Median (Full Range); unit: percent increase in sestamibi AUC
Arm/Group | All Patients Who Received Docetaxel and Tariquidar
Number analyzed (Participants) | 35
percent increase in sestamibi AUC | 82.2 [5.8 to 252]

6. Secondary Outcome: Percent Increase in Sestamibi Area Under Curve (AUC) in Tumor Tissue
Description: 99mTc-sestamibi is a radionuclide imaging agent used to study cardiac function that has also been shown to be a substrate for P-glycoprotein- mediated drug efflux. Because of the high expression of Pgp in liver tissue, sestamibi uptake in liver tissue is often monitored as a marker of Pgp inhibition. A significant change in the area under the curve(AUC) in liver tissue (normal tissue as a surrogate) is defined as P<0.001.
Time Frame: 3-24 hours
Measure: Median (Full Range); unit: Percent
Arm/Group | All Patients Who Received Docetaxel and Tariquidar
Number analyzed (Participants) | 31
Percent | 12.4 [7.2 to 24.1]

ADVERSE EVENTS:
Time Frame: 4 years and 11 months
Arm/Group | Patients on Docetaxel on Days 1, 8 & Tariquidar on Day 8, 22 | Patients on Docetaxel on Days 1, 8 & Tariquidar on Days 1, 22
Serious Adverse Events (participants affected / at risk) | 6/23 | 8/25
Other Adverse Events (participants affected / at risk) | 23/23 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients on Docetaxel on Days 1, 8 & Tariquidar on Day 8, 22 (N=23) | Patients on Docetaxel on Days 1, 8 & Tariquidar on Days 1, 22 (N=25)
BLOOD/BONE MARROW:: Leukocytes (total WBC) (Investigations) | 1 (1) | 1 (1)
CONSTITUTIONAL SYMPTOMS:: Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1) | 0 (0)
CONSTITUTIONAL SYMPTOMS:: (General disorders) | 1 (1) | 2 (2) — Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L)
CONSTITUTIONAL SYMPTOMS:: Rigors, chills (General disorders) | 1 (1) | 0 (0)
DERMATOLOGY/SKIN:: Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL:: Musculoskeletal-Other (Specify,musculoskeletal-lethargic) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NEUROLOGY:: Dizziness/lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
PULMONARY:: Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
PULMONARY:: Pulmonary-Other (Specify,clinical deterioration) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BLOOD/BONE MARROW:: Neutrophils/granulocytes (ANC/AGC) (Investigations) | 0 (0) | 1 (1)
CARDIOVASCULAR (GENERAL):: Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOVASCULAR (GENERAL):: Thrombosis/embolism (Cardiac disorders) | 0 (0) | 2 (2)
GASTROINTESTINAL:: Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEMORRHAGE:: Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEPATIC:: Alkaline phosphatase (Investigations) | 0 (0) | 1 (1)
HEPATIC:: SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 1 (1)
HEPATIC:: SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 1 (1)
INFECTION/FEBRILE NEUTROPENIA:: Febrile neutropenia (fever of unknown origin without clinically or m (Infections and infestations) | 0 (0) | 1 (1)
METABOLIC/LABORATORY:: Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL:: Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NEUROLOGY:: Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
NEUROLOGY:: Mood alteration-anxiety, agitation (Nervous system disorders) | 0 (0) | 1 (1)
PULMONARY:: Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients on Docetaxel on Days 1, 8 & Tariquidar on Day 8, 22 (N=23) | Patients on Docetaxel on Days 1, 8 & Tariquidar on Days 1, 22 (N=25)
AUDITORY/HEARING:: Middle ear/hearing (Ear and labyrinth disorders) | 1 (1) | 0 (0)
BLOOD/BONE MARROW:: Hemoglobin (Blood and lymphatic system disorders) | 18 (130) | 21 (72)
BLOOD/BONE MARROW:: Leukocytes (total WBC) (Blood and lymphatic system disorders) | 18 (86) | 21 (77)
BLOOD/BONE MARROW:: Lymphopenia (Blood and lymphatic system disorders) | 2 (9) | 4 (21)
BLOOD/BONE MARROW:: Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 19 (62) | 16 (41)
BLOOD/BONE MARROW:: Platelets (Blood and lymphatic system disorders) | 7 (22) | 6 (31)
BLOOD/BONE MARROW:: Transfusion: pRBCs (Blood and lymphatic system disorders) | 3 (5) | 9 (11)
CARDIOVASCULAR (ARRHYTHMIA):: Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOVASCULAR (GENERAL):: Edema (Cardiac disorders) | 7 (18) | 8 (8)
CARDIOVASCULAR (GENERAL):: Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOVASCULAR (GENERAL):: Hypotension (Cardiac disorders) | 2 (2) | 1 (1)
CARDIOVASCULAR (GENERAL):: Phlebitis (superficial) (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOVASCULAR (GENERAL):: Thrombosis/embolism (Cardiac disorders) | 2 (3) | 1 (1)
COAGULATION:: Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 9 (17) | 6 (10)
COAGULATION:: Prothrombin time (PT) (Blood and lymphatic system disorders) | 3 (6) | 4 (13)
CONSTITUTIONAL SYMPTOMS:: Fatigue (lethargy, malaise, asthenia) (General disorders) | 18 (42) | 21 (56)
CONSTITUTIONAL SYMPTOMS:: Fever (in the absence of neutropenia, where neutropenia is defined as AGC< (General disorders) | 6 (13) | 4 (5)
CONSTITUTIONAL SYMPTOMS:: Rigors, chills (General disorders) | 1 (1) | 0 (0)
CONSTITUTIONAL SYMPTOMS:: Weight loss (General disorders) | 3 (3) | 3 (3)
DERMATOLOGY/SKIN:: Alopecia (Skin and subcutaneous tissue disorders) | 8 (9) | 8 (10)
DERMATOLOGY/SKIN:: Dermatology/Skin-Other (Specify,_____) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — dermatology/skin: red peeling skin-face
DERMATOLOGY/SKIN:: Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
DERMATOLOGY/SKIN:: Erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DERMATOLOGY/SKIN:: Flushing (Skin and subcutaneous tissue disorders) | 4 (7) | 1 (2)
DERMATOLOGY/SKIN:: Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3)
DERMATOLOGY/SKIN:: Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
DERMATOLOGY/SKIN:: Nail changes (Skin and subcutaneous tissue disorders) | 6 (9) | 8 (8)
DERMATOLOGY/SKIN:: Radiation dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY/SKIN:: Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (4)
GASTROINTESTINAL:: Anorexia (Gastrointestinal disorders) | 12 (21) | 13 (21)
GASTROINTESTINAL:: Constipation (Gastrointestinal disorders) | 10 (13) | 4 (5)
GASTROINTESTINAL:: Dehydration (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL:: Diarrhea patients without colostomy (Gastrointestinal disorders) | 17 (33) | 17 (37)
GASTROINTESTINAL:: Dyspepsia/heartburn (Gastrointestinal disorders) | 3 (5) | 2 (2)
GASTROINTESTINAL:: Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL:: Flatulence (Gastrointestinal disorders) | 1 (1) | 3 (3)
GASTROINTESTINAL:: Gastrointestinal-Other (Specify,_____) (Gastrointestinal disorders) | 1 (1) | 0 (0) — gastrointestinal: tooth fracture
GASTROINTESTINAL:: Mouth dryness (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL:: Nausea (Gastrointestinal disorders) | 13 (34) | 12 (19)
GASTROINTESTINAL:: Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 7 (18) | 8 (13)
GASTROINTESTINAL:: Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 6 (11) | 10 (17)
GASTROINTESTINAL:: Vomiting (Gastrointestinal disorders) | 10 (17) | 7 (8)
HEMORRHAGE:: Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
HEPATIC:: Alkaline phosphatase (Investigations) | 7 (13) | 2 (2)
HEPATIC:: Bilirubin (Investigations) | 5 (14) | 3 (7)
HEPATIC:: Hypoalbuminemia (Metabolism and nutrition disorders) | 16 (36) | 12 (40)
HEPATIC:: SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 7 (11) | 1 (1)
HEPATIC:: SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 5 (6) | 2 (2)
INFECTION/FEBRILE NEUTROPENIA:: Catheter-related infection (Infections and infestations) | 1 (1) | 0 (0)
INFECTION/FEBRILE NEUTROPENIA:: (Infections and infestations) | 3 (3) | 2 (2) — Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0x10e9/L, fever >=38.5 degrees C)
INFECTION/FEBRILE NEUTROPENIA:: (Infections and infestations) | 1 (1) | 1 (1) — Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L)
INFECTION/FEBRILE NEUTROPENIA:: Infection without neutropenia (Infections and infestations) | 4 (7) | 5 (6)
METABOLIC/LABORATORY:: Bicarbonate (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
METABOLIC/LABORATORY:: CPK (creatine phosphokinase) (Investigations) | 1 (1) | 1 (1)
METABOLIC/LABORATORY:: Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
METABOLIC/LABORATORY:: Hyperglycemia (Metabolism and nutrition disorders) | 10 (26) | 11 (23)
METABOLIC/LABORATORY:: Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 3 (5)
METABOLIC/LABORATORY:: Hypermagnesemia (Metabolism and nutrition disorders) | 3 (5) | 3 (4)
METABOLIC/LABORATORY:: Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
METABOLIC/LABORATORY:: Hypocalcemia (Metabolism and nutrition disorders) | 7 (20) | 7 (21)
METABOLIC/LABORATORY:: Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
METABOLIC/LABORATORY:: Hypomagnesemia (Metabolism and nutrition disorders) | 8 (18) | 4 (6)
METABOLIC/LABORATORY:: Hyponatremia (Metabolism and nutrition disorders) | 14 (36) | 15 (26)
METABOLIC/LABORATORY:: Hypophosphatemia (Metabolism and nutrition disorders) | 3 (9) | 1 (1)
MUSCULOSKELETAL:: Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (7)
NEUROLOGY:: Ataxia (incoordination) (Nervous system disorders) | 1 (1) | 0 (0)
NEUROLOGY:: Confusion (Nervous system disorders) | 1 (2) | 1 (1)
NEUROLOGY:: Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
NEUROLOGY:: Dizziness/lightheadedness (Nervous system disorders) | 5 (5) | 3 (3)
NEUROLOGY:: Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1) | 0 (0)
NEUROLOGY:: Insomnia (Nervous system disorders) | 4 (4) | 3 (3)
NEUROLOGY:: Mood alteration-depression (Nervous system disorders) | 2 (2) | 2 (2)
METABOLIC/LABORATORY:: Hypokalemia (Metabolism and nutrition disorders) | 5 (6) | 3 (6)
NEUROLOGY:: Neuropathy-sensory (Nervous system disorders) | 6 (7) | 8 (11)
NEUROLOGY:: Seizure(s) (Nervous system disorders) | 1 (1) | 0 (0)
NEUROLOGY:: Syncope (fainting (Nervous system disorders) | 1 (1) | 0 (0)
NEUROLOGY:: Vertigo (Nervous system disorders) | 1 (1) | 0 (0)
OCULAR/VISUAL:: Conjunctivitis (Eye disorders) | 2 (2) | 0 (0)
OCULAR/VISUAL:: Dry eye (Eye disorders) | 1 (1) | 0 (0)
OCULAR/VISUAL:: Tearing (watery eyes) (Eye disorders) | 9 (11) | 6 (10)
PAIN:: Abdominal pain or cramping (Reproductive system and breast disorders) | 5 (5) | 6 (8)
PAIN:: Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 6 (9) | 6 (10)
PAIN:: Bone pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (5)
PAIN:: Chest pain (non-cardiac and non-pleuritic) (General disorders) | 4 (4) | 0 (0)
PAIN:: Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 7 (22) | 8 (12)
PAIN:: Neuropathic pain (e.g., jaw pain, neurologic pain, phantom limb pain, post-infectious neuralg (Nervous system disorders) | 1 (1) | 0 (0)
PAIN:: Pain-Other (Specify,___) (Nervous system disorders) | 9 (11) | 2 (2) — Back pain Hips + Legs pain-lumbar pain: back pain pain: sore throat pain: chest tube site pain: L flank lower pain: lower back pain pain: lower back
PULMONARY:: Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (3)
PULMONARY:: Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 7 (9)
PULMONARY:: Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (5)
PULMONARY:: Pulmonary-Other (Specify,___) (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) — pleural effusion (malignant)
PULMONARY:: Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RENAL/GENITOURINARY:: Creatinine (Renal and urinary disorders) | 2 (2) | 2 (3)
PULMONARY:: Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
RENAL/GENITOURINARY:: Urinary frequency/urgency (Renal and urinary disorders) | 2 (2) | 1 (1)
ALLERGY/IMMUNOLOGY:: Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 2 (3)
ALLERGY/IMMUNOLOGY:: Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 8 (9) | 3 (3)
PAIN:: Headache (Nervous system disorders) | 5 (5) | 5 (6)
ALLERGY/IMMUNOLOGY:: Allergy-Other (Specify,_____) (Immune system disorders) | 0 (0) | 1 (1) — allergy:reaction to tariquidar
BLOOD/BONE MARROW:: Hemoglobin (Investigations) | 0 (0) | 20 (72)
CARDIOVASCULAR (ARRHYTHMIA):: Palpitations (Cardiac disorders) | 0 (0) | 1 (2)
DERMATOLOGY/SKIN:: Bruising (in absence of grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY/SKIN:: Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
DERMATOLOGY/SKIN:: Wound-non-infectious (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL:: Mucositis due to radiation (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL:: Nausea (Gastrointestinal disorders) | 0 (0) | 12 (19)
HEMORRHAGE:: CNS hemorrhage/bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HEMORRHAGE:: Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 1 (2)
HEMORRHAGE:: Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
INFECTION/FEBRILE NEUTROPENIA:: Infection/Febrile Neutropenia-Other (Specify,____) (Infections and infestations) | 0 (0) | 1 (1) — infection-thrush
METABOLIC/LABORATORY:: Hyperuricemia (Investigations) | 1 (1) | 2 (3)
NEUROLOGY:: Mood alteration-anxiety, agitation (Nervous system disorders) | 0 (0) | 1 (1)
OCULAR/VISUAL:: Ocular/Visual-Other (Specify,___) (Eye disorders) | 0 (0) | 1 (1) — uveitis
OCULAR/VISUAL:: Vision-blurred vision (Eye disorders) | 0 (0) | 2 (2)
PAIN:: Earache (otalgia) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
PAIN:: Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
RENAL/GENITOURINARY:: Dysuria (painful urination) (Renal and urinary disorders) | 0 (0) | 2 (2)
RENAL/GENITOURINARY:: Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No